CLINICAL TRIAL: NCT04795505
Title: Effect of Tertiary A-level Hospital Remote Intervention on MACCE, Adherence to Drugs and Risk Factors Control in Patients With Stable Coronary Artery Disease Compared With Traditional Community Hospital Follow-up
Acronym: CHIPCHAT
Status: Completed | Type: Observational
Sponsor: Chinese Academy of Medical Sciences, Fuwai Hospital (Other)
Responsible Party: Principal Investigator, Weihua Song, Clinical Professor, Chinese Academy of Medical Sciences, Fuwai Hospital
Other Study IDs: CHIPCHAT
Record Dates: First submitted 2021-03-09; First posted 2021-03-12 (Actual); Last update posted 2023-02-16 (Actual); Status verified 2023-02

CONDITIONS: Stable Chronic Angina; Ischemic Heart Disease; Acute Coronary Syndrome
MeSH Terms: conditions — Angina, Stable; Myocardial Ischemia; Acute Coronary Syndrome | interventions — Methods

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Intervention group: A tertiary A-level hospital WeChat-based intervention
  Interventions: Behavioral: Intervention
- Control group: Traditional community hospital intervention
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Intervention — The subsequent visit was through WeChat-based online consultations. Follow-up, assessments and feedback were done at each visit. After follow-up, medication adherence and risk factor modification status were assessed, then individualized feedback, encouragement and recommendations were provided.
  Groups: Intervention group
Behavioral: Control — The subsequent visit was through an offline outpatient clinic at 4 different community hospitals. Participants in this group received standard outpatient cardiology follow-up with formal cardiac rehabilitation and secondary prevention
  Groups: Control group

SUMMARY:
The study was a multicenter, two-arm, parallel, open label, prospective study intended for to compare effect of offline community hospital intervention on adherence to drugs and risk factors control in patients with stable coronary artery disease compared with tertiary A-level hospital WeChat-based intervention.

DETAILED DESCRIPTION:
Objective: This study is intended for to compare effect of offline community hospital intervention on adherence to drugs and risk factors control in patients with stable coronary artery disease compared with tertiary A-level hospital WeChat-based intervention.

Study design: The study was a multicenter, two-arm, parallel, open label, prospective study that evaluated a WeChat-based intervention offered by tertiary A-level hospital with 1 year of follow-up.

Study intervention: All patients received lifestyle intervention and drug adjustment at 1 month, 3 months, 6 months and 1 year follow-up. In the control group, the subsequent visit was through an offline outpatient clinic at 4 different community hospitals. Participants in this group received standard outpatient cardiology follow-up with formal cardiac rehabilitation and secondary prevention. While in the intervention group, the subsequent visit was through WeChat-based online consultations.

Outcome measures: The primary outcome was MACCE. Secondary outcome included blood pressure, heart rates, smoking cessation, drinking cessation, body mass index, and medications adherence.

Statistical analysis: Values of analyzed endpoints between intervention group and control group will be compared according to the analysis plan. We'll follow a prespecified analysis plan and subgroup analysis will be conducted accordingly.

ELIGIBILITY:
Inclusion Criteria:

1. aged between 18-99 years
2. diagnosed with SCAD according to guidelines by coronary CTA or coronary angiography (including stable angina, ischemic cardiomyopathy, and the stable course after acute coronary syndrome)
3. have sufficient Chinese language proficiency to reading, speaking and listening
4. live with at least one caregiver or guardian in the household
5. presence of stable hemodynamics without using vasopressor
6. able to individually consent
7. not participating in any other clinical trial

Exclusion Criteria:

1. unable to provide informed consent
2. unable to be involved in clinical follow up and treatment
3. suffered comorbidity with a life expectancy of less than 1 year
4. have contra-indication to cardiac rehabilitation
5. acute coronary syndrome

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants are screened from several community hospitals and tertiary-A hospitals in Beijing
Sampling Method: Non-Probability Sample
Enrollment: 1424 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-01-01 (Actual)

PRIMARY OUTCOMES:
MACCE | 1 year
  acute myocardial infarction, acute heart failure, stroke, rehospitalization for cardiovascular event, death from a cardiovascular cause and unplanned revascularization

SECONDARY OUTCOMES:
blood pressure | 1 year
  BP was measured twice by an electronic device after 10 min of seated rest and calculated as the mean of 2 measurements.
heart rates | 1 year
  standard protocol
smoking cessation | 1 year
  self-reported
drinking cessation | 1 year
  self-reported
body mass index | 1 year
  standard protocol
medications adherence | 1 year
  self-reported
LDL | 1 year
  standard protocol
HbA1c | 1 year
  standard protocol

CONTACTS AND LOCATIONS:
Overall Officials: Weihua Song, MD, Principal Investigator — Fuwai Hospital, Chinese Academy of Medical Science; National Center for Cardiovascular Diseases
Locations (1):
- Fuwai Hospital, Chinese Academy of Medical Science; National Center for Cardiovascular Diseases, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zheng X, Spatz ES, Bai X, Huo X, Ding Q, Horak P, Wu X, Guan W, Chow CK, Yan X, Sun Y, Wang X, Zhang H, Liu J, Li J, Li X, Spertus JA, Masoudi FA, Krumholz HM. Effect of Text Messaging on Risk Factor Management in Patients With Coronary Heart Disease: The CHAT Randomized Clinical Trial. Circ Cardiovasc Qual Outcomes. 2019 Apr;12(4):e005616. doi: 10.1161/CIRCOUTCOMES.119.005616. PMID 30998400
- [Background] Yu C, Liu C, Du J, Liu H, Zhang H, Zhao Y, Yang L, Li X, Li J, Wang J, Wang H, Liu Z, Rao C, Zheng Z; MISSION-2 Collaborative Group. Smartphone-based application to improve medication adherence in patients after surgical coronary revascularization. Am Heart J. 2020 Oct;228:17-26. doi: 10.1016/j.ahj.2020.06.019. Epub 2020 Jul 4. PMID 32745732
- [Background] Chen X, Zhou X, Li H, Li J, Jiang H. The value of WeChat application in chronic diseases management in China. Comput Methods Programs Biomed. 2020 Nov;196:105710. doi: 10.1016/j.cmpb.2020.105710. Epub 2020 Aug 14. PMID 32858284
- [Derived] Shi B, Liu X, Dong Q, Yang Y, Cai Z, Wang H, Yin D, Wang H, Dou K, Song W. The Effect of a WeChat-Based Tertiary A-Level Hospital Intervention on Medication Adherence and Risk Factor Control in Patients With Stable Coronary Artery Disease: Multicenter Prospective Study. JMIR Mhealth Uhealth. 2021 Oct 27;9(10):e32548. doi: 10.2196/32548. PMID 34569467
- See also: Number of monthly active WeChat users from 2nd quarter 2011 to 2nd quarter 2020(in millions) — https://www.statista.com/statistics/255778/number-of-active-wechat-messenger-accounts/#statisticContainer